0453-01-01/

# STATISTICAL ANALYSIS PLAN

A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.05% to TAZORAC® (tazarotene) Cream 0.05% and Both Active Treatments to a Vehicle Control in the Treatment of Stable Plaque Psoriasis

Protocol Number: 0453-01-01 / NCT02886702

# **Sponsor:**

Fougera Pharmaceuticals Inc. 60 Baylis Road Melville, New York, 11747

**Contract Research Organization:** 

April 26, 2017

Final Version 2.0

**Tazarotene Cream 0.05%** 

Protocol /

0453-01-01/

# SAP FINAL VERSION APPROVALS

A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study Comparing Tazarotene Cream 0.05% to TAZORAC® (tazarotene) Cream 0.05% and Both Active Treatments to a Vehicle Control in the Treatment of Stable Plaque Psoriasis

| Written By: | |
|--------------|-------|
| Signature: | Date: |
| Reviewed By: | |
| Reviewed By. | |
| Signature: | Date: |
| Approved By: | |
| Signature: | Date: |

Tazarotene Cream 0.05% Protocol / 0453-01-01/

**Revision History** 

Tazarotene Cream 0.05%

Protocol /

0453-01-01/

### List of Abbreviations and Definition of Terms

ADaM Analysis Data Model

AE Adverse Event

ANOVA Analysis of Variance BSA Body Surface Area

C Celsius

CDISC Clinical Data Interchange Standards Consortium

CI Confidence Interval CRF Case Report Form

CRO Contract Research Organization eCRF Electronic Case Report Form

EOS End of Study Early Termination

F Fahrenheit

FDA Food and Drug Administration

Hg Mercury

ICF Informed Consent Form

ICH International Conference on Harmonisation

IGA Investigator Global Assessment

IP Investigational Product

LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

mITT modified Intent-to-Treat Population

OGD Office of Generic Drugs
PASI Psoriasis Area Severity Index

PD Protocol Deviation

PP Per-Protocol

RLD Reference Listed Drug
SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System

SD Standard Deviation

SDTM Study Data Tabulation Model

# TABLE OF CONTENTS

| 1. INTRODUCTION |
|---|
| 2. OBJECTIVES |
| 3. OVERALL STUDY DESIGN7 |
| 4. RANDOMIZATION AND BLINDING11 |
| 5. SAMPLE SIZE |
| 6. ANALYSIS POPULATION12 |
| 7. STUDY EFFICACY VARIABLES |
| 8. STATISTICAL ANALYSIS METHODS |
| 8.1 Baseline Characteristics |
| 8.1.1 Demographics Comparability of Treatment Groups |
| 8.1.2 Medical History |
| 8.1.3 Concomitant Medications |
| 8.1.4 Pregnancy Test |
| 8.2 Primary and Secondary Endpoint Analyses |
| 8.3 Safety Analysis |
| 8.3.1 Adverse Events |
| 8.3.2 Application Site Reactions |
| 8.3.3 Vital Signs |
| 8.4 Multiple Comparisons |
| 8.5 Methods for Handling Missing Data |
| 8.6 Interim Analyses |
| 9. TABLE, LISTING AND FIGURE SHELLS19 |
| T16.1.9.1 Summary of Discontinued Subjects (Safety Population) |
| T16.1.9.2 Summary of Protocol Deviations_(Safety Population) |
| T16.1.9.3.1 Summary of Subjects Excluded from Efficacy Analysis |
| T16.1.9.3.2 Summary of Subjects Included in Analysis Population by Study Center 24 |
| T16.1.9.4.1 Summary of Demographic Data (Safety Population) |
| T16.1.9.4.2 Summary of Baseline Parameters (Safety Population) |
| T16.1.9.5.1 Summary of Demographic Data (modified Intent-to-Treat Population)29 |
| T16.1.9.5.2 Summary of Baseline Parameters (modified Intent-to-Treat Population) 29 |
| T16.1.9.6.1 Summary of Demographic Data (Per-Protocol Population) |
| T16.1.9.6.2 Summary of Baseline Parameters (Per-Protocol Population) |
| T16.1.9.7.1 Summary of Analysis Results of Primary Efficacy Endpoint |
| T16.1.9.7.2 Summary of Supportive Analysis Results of Primary Efficacy Endpoint 31 |
| T16.1.9.8.1 Summary of Analysis Results of Secondary Efficacy Endpoint |
| T16.1.9.8.2 Summary of Supportive Analysis Results of Secondary Efficacy Endpoint |
| Proportion of Subjects with Disease Severity (a score of 0 or 1) on IGA at the Week 12 |
| Visit |
| T16.1.9.9.1 Summary of Analysis Results of Secondary Efficacy Endpoint |

| Tazarotene Cream 0.05% | Protocol / | 0453-01-01/ |
|---|---|---|
| T16.1.9.9.2 Summary of Supportive Analys | is Results of Secondary E | fficacy Endpoint 35 |
| T16.1.9.10 Overall Summary of Adverse Ev | • | • • |
| T16.1.9.11 Summary of Frequency of All A | | |
| T16.1.9.12 Summary of Frequency for AEs | Occurring in at Least 5% | of Subjects by Body |
| System (Safety Population) | ••••• | 37 |
| T16.1.9.13 Summary of Frequency of All A | dverse Events by Severity | (Safety Population)38 |
| T16.1.9.14 Summary of Frequency of All A | dverse Events by Relation | nship (Safety Population) |
| | | 39 |
| T16.1.9.15 Summary of Frequency of Serio | us Adverse Events (Safet | y Population)40 |
| T16.1.9.16 Summary of Application Site Re | eaction (Safety Population | n)41 |
| T16.1.9.17 Summary of Frequency of Appl | ication Site Reaction (Saf | ety Population) 42 |
| T16.1.9.18 Summary of Vital Signs (Safety | / Population) | 43 |
| L16.2.1 Listing of Discontinued Subjects | | |
| L16.2.2 Listing of Protocol Deviations | | 45 |
| L16.2.3.1 Subjects Excluded from the Per-P | | |
| L16.2.3.2 Subjects Excluded from the Modi | | |
| L16.2.4.1 Listing of Demographic Data | | |
| L16.2.4.2 Listing of Medical History | | |
| L16.2.4.3 Listing of Concomitant Medication | | |
| L16.2.5.1 Listing of Visit Date Information | | 51 |
| L16.2.5.2 Listing of Drug Administration | | |
| L16.2.6.1 Listing of Investigator Global Ass | | |
| L16.2.6.2 Listing of Psoriasis Area Severity | | |
| L16.2.6.3 Listing of Dermatological Examin | | |
| L16.2.7.1 Listing of Adverse Events by Tre | | |
| L16.2.7.2 Listing of Application Site Reacti | | |
| L16.2.8.1 Listing of Pregnancy Test Results | | |
| L16.2.8.2 Listing of Vital Signs | | |
| APPENDIX A: Investigator's Global Asses | | |
| APPENDIX B: Psoriasis Area Severity Inde | | |
| APPENDIX C: Application Site Reactions. | | 62 |

**Tazarotene Cream 0.05%** 

Protocol /

0453-01-01/

### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol 0453-01-01 Rev. 2 dated 12/22/2016. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol 0453-01-01 Rev. 2 dated 12/22/2016
- Final eCRF Version 1.0 for

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a subject in this study.

# 2. OBJECTIVES

The objectives of this study are to:

- 1. Evaluate the therapeutic equivalence of the Test product, Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) to the Reference product, TAZORAC® (tazarotene) Cream 0.05% (Allergan, Inc.) in the treatment of stable plaque psoriasis.
- 2. Demonstrate the superiority of the efficacy of the Test and Reference (active) products over that of the Placebo in the treatment of stable plaque psoriasis.
- 3. Compare the safety of the Test, Reference and Placebo products in the treatment of stable plaque psoriasis.

# 3. OVERALL STUDY DESIGN

This multi-center, double-blind, randomized, vehicle-controlled, parallel-group, bioequivalence clinical study has been designed to evaluate the efficacy and safety of a

# Tazarotene Cream 0.05%

Protocol /

0453-01-01/

generic tazarotene cream 0.05% (Fougera Pharmaceuticals Inc.) compared to the FDA Reference Listed Drug (RLD) TAZORAC® (tazarotene) Cream 0.05% (Allergan) in subjects with a clinical diagnosis of stable plaque psoriasis of at least moderate severity. Additionally, both the Test product and Reference (i.e., the RLD) products will be tested for superiority to a Placebo. Subjects with confirmed stable plaque psoriasis will apply the investigational product (IP) once daily, in the evening, to psoriatic lesions for  $84 \pm 4$  days (12 weeks).

Before any study-specific procedures are performed, all subjects will read and sign the IRB-approved ICF.

Each site will develop an individualized recruitment plan to collectively enroll approximately 855 eligible subjects, 18 years of age and older, with a clinical diagnosis of stable plaque psoriasis and meeting the inclusion/exclusion criteria. Subjects will be randomized to one of the three IPs as follows:

- Test: Tazarotene Cream, 0.05% (Fougera Pharmaceuticals Inc.)
- Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)
- Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Subjects will attend the following scheduled clinic visits:

- Visit 1 Screening/Baseline: Day -14 to Day 1
- Visit 2 Interim Visit: Day  $28 \pm 4$  days
- Visit 3 Interim Visit: Day  $56 \pm 4$  days
- Visit 4 End of Study: Day  $85 \pm 4$  days

Subjects may attend unscheduled clinic visits:

• Visit 9999 – Unscheduled visit

At Visit 1, eligible subjects will be randomized to the Test, Reference or Placebo product in a 1:1:1 ratio using the system, which is an interactive response technology (IRT) system provided by the IRT provider. Study subjects will be provided with may be dispensed to the subject at the discretion of the Investigator if the subject has a high BSA affected with plaque psoriasis at the time of dispensation that would warrant additional product. At Visit 2 and Visit 3, subjects who continue to be eligible for continuation in the study can be dispensed an additional of IP, as needed based on the subject's current BSA affected and the amount of IP remaining from the tube(s) previously dispensed. Further, any empty tubes will be collected at these visits. At Visit 4, all tubes will be collected (used and unused). A subject may return for an Unscheduled Visit at any time, should they require a resupply of IP (i.e., tube lost; all IP used between visits). It is estimated that approximately , but up to may be needed to dose a subject with

Tazarotene Cream 0.05%

Protocol /

0453-01-01/

high BSA involvement (~20% BSA) for the treatment period (depending upon their treatment response over the 12 weeks). Subjects with less BSA involvement will need significantly less IP (approximately 2 to 4 tubes).

The day that the subject administers their first dose of IP will be considered Day 1.

For all other

subjects, the first dose (Day 1) of IP will be applied on the evening of Visit 1.

The subject will be instructed to apply enough cream  $(2 \text{ mg/cm}^2)$  to cover only the psoriatic lesions with a thin film  $(2 \text{ mg/cm}^2)$  once daily, in the evening, until the evening before Visit 4 (Day  $85 \pm 4$  days). There will be no application of the product on the day of the End of Study visit.

Efficacy evaluations will be based on dermatological assessments in the clinic. The primary statistical analysis of interest is the (1) proportion of subjects with treatment success (defined as none, minimal or mild disease, a score of 0, 1 or 2, within the treatment area) on the Investigator's Global Assessment (IGA) at the Week 12 visit. The secondary analyses are (1) proportion of subjects with disease severity at the Week 12 visit consistent with none or minimal, a score of 0 or 1, within the treatment area on the IGA, and (2) proportion of subjects with target site plaque elevation, scaling, and erythema scores of less than or equal to one on the PASI at the Week 12 visit. PASI is the sum of the three individual component scores.

**Tazarotene Cream 0.05%** 

Protocol /

0453-01-01/

# **Study Schematic**

| PROCEDURE | VISIT 1<br>(Day -14 to<br>1)<br>Screening/<br>Baseline | VISIT 2<br>(Day 28<br>± 4 Days)<br>Interim Visit | VISIT 3<br>(Day 56<br>± 4 Days)<br>Interim Visit | VISIT 4 (Day 85 ± 4 Days)* End of Study/ Early Termination |
|---|---|---|---|---|
| Informed Consent | X <sup>‡</sup> | | | |
| Medical History/ | X <sup>‡</sup> | | | |
| Demographics | | | | |
| Pregnancy Test <sup>†</sup> | $X^{\ddagger}$ | X | X | X |
| Vital Signs | $\mathbf{X}^{\ddagger}$ | | | X |
| Dermatologic Assessment | X‡ | | | |
| IGA | X‡ | X | X | X |
| PASI Assessment | X <sup>‡</sup> | X | X | X |
| Application Site Reactions | X | X | X | X |
| Inclusion/Exclusion Criteria<br>Review | X <sup>‡</sup> | | | |
| Concomitant Medication | X <sup>‡</sup> | X | X | X |
| Randomization | X | | | |
| Dispense IP | X | X** | X** | |
| Return of IP | | X** | X** | X |
| Dispense Subject Diary/Supplies | X | X | X | |
| Collect/Review Subject Diary | | X | X | X |
| Adverse Events | | X | X | X |
| Discharge from Study | | | | X |

<sup>\*</sup> Dosing regimen is once daily in the evening for 84 days (Day 1 to Day 84) through the evening before Visit 4 (Day 85 ± 4)

\*\* If applicable, based on use of previously dispensed product.

† For females of childbearing potential

<sup>&</sup>lt;sup>‡</sup> Procedures performed as part of the screening assessment, before randomization

Tazarotene Cream 0.05% Protocol / 0453-01-01/

### 4. RANDOMIZATION AND BLINDING

| The IP will be randomized, packaged and blinded by an |
|---|
| . The randomization code will be generated using a validated computer |
| program. Each |
| site will receive multiple, full blocks of IP in each delivery. The quantity received may vary. |
| Randomization will be pre-planned according to a computer-generated randomization scheme. The randomization code will be retained within which is maintained by will also retain the kit boxes numbers supplied to each site and the kit boxes numbers that have been selected for retention and are therefore unavailable for dispensing to subjects. |
| Upon confirmation of subject eligibility, the subject's information (i.e., subject's initials, date of birth, etc.) will be entered into and the system will assign a randomization number to the subject based upon subject a kit box number in a blinded fashion at Visit 1. This kit box number will correspond to a specific treatment group within the subject. The site will record the randomization number and the kit box number in the subject's source documentation and drug dispensing log. The will record the tube number of the subject's source documentation and drug dispensing log. At Visits 2, 3 and/or Unscheduled Visit, additional IP may be dispensed to the subject, as needed. The an additional unused tube from the subject's previously assigned kit box, dispense it to the subject and record the tube number. |
| Each subject will |
| maintain the same treatment assignment throughout the study. |

# 5. SAMPLE SIZE

Sample size calculations were performed using endpoint analysis, the rate of treatment success for the Reference treatment after 12 weeks of treatment is expected to be approximately in the PP population. Assuming that the rates of treatment success for Test and Reference treatments are the same, a sample size of subjects in each active group in the PP population will provide approximately power to demonstrate therapeutic equivalence (i.e., the 90% confidence interval (Yates' continuity-corrected) of the absolute difference between the Test and Reference rates of treatment success is within a defined equivalence range [-20% to + 20%]).

| 1 azarotene Cream 0.05% | Protocol / | 0453-01-01/ |
|---|---|---|
| The rates of treatment success for the Placebot treatment are assumed to be approximately population. Using a 1:1 (active: placebo) rand rate from mITT to PP population will be about Reference and Placebo) of the mITT population superiority of active over Placebo at the 5% sit corrected Z-Tests and a pooled response raproportions). | and at least omization scheme, subjects in will provide at least gnificance level (p | respectively, in the mITT and assuming the conversion in each treatment group (Test, ast power to demonstrate < 0.05, two-sided continuity- |
| Under the above assumptions, the overall stude and superiority is estimated to be at least may drop out from the study or are otherw randomized to obtain subjects in the mITT | To allow for approxise non-evaluable, | of subjects who up to 855 subjects may be |
| 6. ANALYSIS POPULATION | | |
| Per-Protocol Population | | |
| The PP population will include subjects that con | nply with the protoc | col as follows: |
| <ul> <li>All randomized subjects who meet all in</li> <li>Make the final study visit (Visit 4) with no PDs that would affect the integrity of</li> <li>Comply with study restrictions including</li> <li>Apply the IP appropriately and are with 12 weeks (Day 85 ± 4) of treatment.</li> <li>Do not miss the scheduled applications in</li> </ul> | tin the protocol win the data. g concomitant medication com | dow of Day $85 \pm 4$ days with |

**Tazarotene Cream 0.05%** 

Protocol /

0453-01-01/

# **Modified Intent-to-Treat Population (mITT) Population**

The mITT population will include all subjects in the PP population plus all randomized subjects who meet all inclusion/exclusion criteria, apply at least one dose of assigned product, and return for at least one post-Baseline evaluation.



# **Safety Population**

All subjects who are randomized and received IP will be included in the analysis of safety.

### 7. STUDY EFFICACY VARIABLES

# **Primary Efficacy Endpoints**

Proportion of subjects with treatment success (defined as none, minimal or mild disease, a score of 0, 1 or 2 within the treatment area) on the IGA at the Week 12 visit (Day  $85 \pm 4$  days, End of Study).

# **Secondary Efficacy Endpoints**

1. Proportion of subjects with disease severity at the Week 12 visit (Day  $85 \pm 4$  days, End of Study) consistent with none or minimal, a score of 0 or 1, within the treatment area on the IGA

# AND

2. Proportion of subjects with target site plaque elevation, scaling and erythema scores of less than or equal to 1 on the PASI at the Week 12 visit (Day  $85 \pm 4$ , End of Study).

# 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p<0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics, efficacy variables and safety variables.

For categorical variables, the number and percent of each category within a parameter will be

Tazarotene Cream 0.05%

Protocol /

0453-01-01/

calculated for non-missing data. For continuous variables with non-missing values, statistics will include number of observations, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS®, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model).

### 8.1 Baseline Characteristics

# 8.1.1 Demographics Comparability of Treatment Groups

Baseline characteristics will be evaluated separately for the PP, mITT and Safety populations.

Demographic information collected at baseline includes the following:

- Age (years)
- Sex (Male/Female)
- Ethnicity (Hispanic/non Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)
- Baseline total BSA affected with Psoriasis
- Baseline percent BSA affected with Psoriasis
- Baseline PASI Score (the sum of the three individual component scores)
- Baseline Scores for Individual Components (Erythema, Scaling and Plaque Elevation)
- Baseline IGA Score
- Treatment location
- Treatment area size (area)
- Target lesion size (area)

Summary tables by treatment group will be presented. Continuous variables will be summarized using descriptive statistics (number of observations, median, minimum, maximum, mean and standard deviation). Categorical variables will be summarized using frequencies and percentage. Baseline treatment comparisons will be presented using Chi-Square test for the categorical variables, and Analysis of Variance (ANOVA) for the continuous variables.

All data will be listed by treatment and subject.

Tazarotene Cream 0.05%

Protocol /

0453-01-01/

# **8.1.2** Medical History

At Visit 1 subjects will be questioned about their personal medical history, including psoriasis history. The medical history will include a complete review of all current diseases and their respective durations and treatments.

Medical history data will be listed by treatment and subject.

## **8.1.3 Concomitant Medications**

At Visit 1, subjects will be questioned about current and prior concomitant medication use over the 6 months. Subjects will also be questioned about ongoing or new concomitant medication use during the treatment period at Visits 2, 3 and 4.

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment and subject.

# 8.1.4 Pregnancy Test

All females of childbearing potential will have a urine pregnancy test performed at each Scheduled visit. All females of childbearing potential will have a urine pregnancy test performed at Visit 1 (Baseline), Visit 2, Visit 3, and Visit 4 (or early termination).

Pregnancy test results will be listed by treatment and subject.

# 8.2 Primary and Secondary Endpoint Analyses

# **Therapeutic Bioequivalence Analysis**

Therapeutic equivalence will be evaluated for both primary and secondary endpoints using the PP population, with results in the mITT population being supportive.

Based on the usual method used in OGD for binary outcomes, the 90% confidence interval for the difference in success proportions between test and reference treatment should be contained within [-0.20, +0.20] in order to establish equivalence.

The compound hypothesis to be tested is:

$$H_0: P_T - P_R < -.20 \text{ or } P_T - P_R > .20 \text{ versus}$$

# Tazarotene Cream 0.05%

Protocol /

0453-01-01/

$$H_A: -.20 \le P_T - P_R \le .20$$

where  $P_T$  = success rate of test treatment

 $P_R$  = success rate of reference treatment.

Let

 $n_T$  = sample size of test treatment group

 $cn_T$  = number of patients considered as Treatment Success in test treatment group

 $n_R$  = sample size of reference treatment group

 $cn_R$  = number of patients considered as Treatment Success in reference treatment group

$$\hat{P}_T = c n_T / n_T$$
  $\hat{P}_R = c n_R / n_R$ , and

$$se = (\widehat{P}_T (1 - \widehat{P}_T)/n_T + (\widehat{P}_R (1 - \widehat{P}_R)/n_R)^{1/2})$$

The 90% confidence interval for the difference in proportions between test and reference will be calculated as follows, using Yates' correction:

$$L = (\hat{P}_T - \hat{P}_R) - 1.645 se - (1/n_T + 1/n_R)/2$$

$$U = (\hat{P}_T - \hat{P}_R) + 1.645 se + (1/n_T + 1/n_R)/2$$

For the proportion of Treatment Success, if the 90% confidence interval (with Yates' Correction Factor) of the difference between the proportion of subjects considered a "treatment success" in the Test and the Reference treatment groups at Week 12 is contained within the pre-defined equivalence limits [-20%, +20%], then therapeutic equivalence will be considered to have been supported for the endpoint. The same statistical approach will be conducted for analysis of the two dichotomized secondary endpoints in the PP and mITT populations.

To declare therapeutic equivalence of the Test product to the Reference product, therapeutic equivalence must be demonstrated for only the primary endpoint in the PP population.

# **Superiority to Placebo Analysis**

The primary measure of superiority will be evaluated using the mITT population and LOCF for missing efficacy values. The results in the PP population will be considered supportive.

The superiority of the Test and Reference products over Placebo will be concluded for the primary endpoint if the proportion of treatment success at Week 12 is statistically superior to Placebo (p < 0.05, two-sided a Cochran-Mantel-Haenszel exact test stratified by clinical site) using the mITT population and LOCF. The same statistical approach will be conducted for analysis of the two dichotomized secondary endpoints in the mITT and PP populations.

Tazarotene Cream 0.05%

Protocol /

0453-01-01/

.

To declare superiority of the Test and Reference products over Placebo, their superiority must be demonstrated for only the primary endpoint in the mITT population.

A summary table with frequency and percentage of the proportion of Treatment Success by treatment group will be presented.

# **Treatment-by-Site Interaction and Pooling of Clinical Sites**

As this is a multiple-site study, the interaction of treatment-by-site may be evaluated by the Cochran-Mantel-Haenszel test (stratified by site) at the 5% significance level (p < 0.05, 2-sided) for the primary efficacy endpoint in both the PP population (for equivalence testing) and mITT population (for superiority testing).

If the treatment-by-site interaction is found to be statistically significant (p < 0.05) then the interaction will also be assessed for clinical relevance before pooling the data across sites. This will include examination of responder rates at each site where sample sizes per treatment may be influential in the assessment of the interaction.

# 8.3 Safety Analysis

All safety analyses will be based on the Safety Population.

# 8.3.1 Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 18.1 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, relationship to the IP, action taken and outcome.

In each of the following categories, the total number and percentage of subjects with 1) at least one AE, 2) discontinued study drug due to AEs, 3) AE severity and AEs related to the IP, 4) serious AEs and death will be summarized separately by treatment groups.

A summary table of the number and percent of subjects with AEs by system organ class, preferred term, and treatment group will be presented. Each subject will be counted only once within each preferred term.

# Tazarotene Cream 0.05%

Protocol /

0453-01-01/

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and treatment group will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to the IP, and treatment group will be presented. Relationship to a study drug will be classified as "Suspected" or "Not Suspected".

Should sufficient data exist, adverse event frequencies will be compared between treatments using Fisher's exact test.

# **8.3.2** Application Site Reactions

At Visits 1, 2, 3 and 4 the Investigator will evaluate the subject for local application site reactions.

Signs and Symptoms recorded at each visit will be compared between treatment groups. Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) comparing the application site reactions for each treatment group will be presented by visit.

A frequency summary table comparing the application site reactions for each treatment group will be presented by visit.

### 8.3.3 Vital Signs

The subject's vital signs (pulse, blood pressure, temperature and respiration rate) will be recorded at Visit 1 and Visit 4.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by treatment and visit for non-missing values.

All data will be listed by treatment and subject.

# 8.4 Multiple Comparisons

No multiple comparison adjustment will be made in this study.

# 8.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available

Tazarotene Cream 0.05%

Protocol /

0453-01-01/

data. Subjects with missing data will be excluded only from analyses for which data are not available, including denominators.

Subjects who discontinue early for reasons besides lack of treatment effect or worsening of condition should be excluded from the PP population, but included in the modified Intent-to-Treat (mITT) population using the last observation carried forward (LOCF), provided they administered at least one dose of randomized IP and completed at least one post-dose evaluation.

# 8.6 Interim Analyses

There is no interim analysis planned in this study.

# 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

| Fougera Pharmaceuticals Inc. | | |
|------------------------------|------------|-------------|
| Tazarotene Cream 0.05% | Protocol / | 0453-01-01/ |

# TABLE, LISTING AND FIGURE SHELLS

T16.1.9.1 Summary of Discontinued Subjects (Safety Population)

| Subjects | Test | Reference | Placebo | Total |
|--------------------------|------|-----------|---------|-------|
| Randomized | XXX | XXX | XXX | xxx |
| Completed Study | XXX | XXX | XXX | xxx |
| Terminated Early | xxx | xxx | xxx | xxx |
| Early Termination Reason | | | | |
| Administrative reasons | xxx | XXX | xxx | XXX |
| Lack of efficacy | xxx | XXX | xxx | XXX |
| Lost to Follow-Up | xxx | xxx | xxx | xxx |
| etc. | | | | |

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

T16.1.9.2 Summary of Protocol Deviations (Safety Population)

| | Test | Reference | Placebo | Total |
|-----------------------------------------|------|-----------|---------|-------|
| Total Subjects with Protocol Deviations | xxx | XXX | xxx | XXX |
| Total Deviations | xxx | XXX | xxx | xxx |
| Lost to follow up | xxx | xxx | xxx | xxx |
| Outside visit window | xxx | xxx | xxx | xxx |
| Missed Visit | XXX | XXX | XXX | XXX |
| Restricted Medication | xxx | xxx | xxx | xxx |
| etc | XXX | XXX | XXX | XXX |
| Other | XXX | xxx | xxx | XXX |

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

Protocol / 0453-01-01/

T16.1.9.3.1 Summary of Subjects Excluded from Efficacy Analysis (Population Determination)

| | | Test | Reference | Placebo | Total |
|---|---|---|---|---|---|
| Randomized | Total | xxx | XXX | XXX | XXX |
| Safety Population | Total | xxx | XXX | xxx | XXX |
| Excluded from Safety | Did not received study product | XXX | xxx | XXX | xxx |
| | etc. | | | | |
| mITT Population | Total | XXX | XXX | XXX | XXX |
| Excluded from mITT | Did not received study product | XXX | XXX | XXX | XXX |
| | etc. | | | | |
| PP Population | Total | xxx | xxx | xxx | XXX |
| Excluded from Excluded from PP | Restricted Medication | XXX | xxx | XXX | xxx |
| | etc. | | | | |

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

Tazarotene Cream 0.05%

Protocol /

0453-01-01/

T16.1.9.3.2 Summary of Subjects Included in Analysis Population by Study Center

| | | | | | PP | | | _ | mITT | | | | Safety | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site<br>No. | Name | Total<br>Randomized | Test | Ref | Placebo | Total | Test | Ref | Placebo | Total | Test | Ref | Placebo | Total |
| XX | XXXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX | XXX | xxx | XXX |
| XX | XXXX | XXX | XXX | xxx | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | xxx |

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\



Created on: ddmmmyy hh:mm

0453-01-01/

T16.1.9.4.1 Summary of Demographic Data (Safety Population)

| | | Test | Reference | Placebo | |
|---|---|---|---|---|---|
| | | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | P-value |
| Age (years) | n | xxx | xxx | xxx | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | xx.x | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Race | White | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Black/African American | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Native Hawaiian or other Pacific Islander | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Asian | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | American Indian or Alaska Native | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Sex | Female | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Male | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Ethnicity | Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Not Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

N= number of subjects in the treatment group; n= number of subjects with data available; % is based on N

P-values are from Chi-squre test for categorical variables and ANOVA for the continuous variables.

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

0453-01-01/

T16.1.9.4.2 Summary of Baseline Parameters (Safety Population)

| | | Test | Reference | Placebo | |
|---|---|---|---|---|---|
| | | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | P-value |
| Total BSA affected with Psoriasis | n | XXX | XXX | XXX | x.xxxx |
| | $\text{Mean} \pm \text{SD}$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Total percent BSA affected with Psoriasis | n | XXX | XXX | XXX | x.xxxx |
| | $\text{Mean} \pm \text{SD}$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Baseline IGA Score | n | XXX | XXX | XXX | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | xx.x | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Baseline PASI Score | n | XXX | XXX | XXX | x.xxxx |
| | $\text{Mean} \pm \text{SD}$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | xx.x | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |

Note: N= number of subjects in the treatment group; n= number of subjects with data available; % is based on N=

P-values are from Chi-squre test for categorical variables and ANOVA for the continuous variables.

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT Created on: ddmmmyy hh:mm Page 2 of N

0453-01-01/

T16.1.9.4.2 Summary of Baseline Parameters (Safety Population)

| | | Test | Reference | Placebo | |
|---|---|---|---|---|---|
| | | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | P-value |
| Erythema | Clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Almost clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Very severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Scaling | Clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Almost clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Very severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| laque Elevation | Clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | X.XXXX |
| | Almost clear | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Very severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

Note: N= number of subjects in the treatment group; n= number of subjects with data available; % is based on N

P-values are from Chi-squre test for categorical variables and ANOVA for the continuous variables.

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Tazarotene Cream 0.05%

Protocol /

0453-01-01/

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

\SAS\OUT

Created on: ddmmmyy hh:mm

Page 3 of N

# **T16.1.9.4.2 Summary of Baseline Parameters** (Safety Population)

| | | Test | Reference | Placebo | _ |
|---|---|---|---|---|---|
| | | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | P-value |
| Treatment area size (area) | n | XXX | XXX | XXX | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | xx.x | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Target lesion size (area) | n | XXX | XXX | xxx | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Treatment location | Head front | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Head back | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Torso front | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Torso back | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | etc | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

Note: N= number of subjects in the treatment group; n= number of subjects with data available;

% is based on N

P-values are from Chi-squre test for categorical variables and ANOVA for the continuous variables.

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\ \SAS\OUT Created on: ddmmmyy hh:mm

Similar tables will be created for T16.1.9.5.1, T16.1.9.5.2, T16.1.9.6.1 and T16.1.9.6.2

T16.1.9.5.1 Summary of Demographic Data (modified Intent-to-Treat Population)

T16.1.9.5.2 Summary of Baseline Parameters (modified Intent-to-Treat Population)

T16.1.9.6.1 Summary of Demographic Data (Per-Protocol Population)

T16.1.9.6.2 Summary of Baseline Parameters (Per-Protocol Population)

0453-01-01/

# T16.1.9.7.1 Summary of Analysis Results of Primary Efficacy Endpoint Proportion of Treatment Successes on the IGA (a score of 0 or 1 or 2) at the Week 12 Visit

| Equivalence: Per-Protocol Population | | | | | |
|---|---|---|---|---|---|
| | Number of | | | Difference Between Treatments | |
| Treatment | | Number of<br>Treatment | Proportion of<br>Treatment | | |
| Group | Subjects (N) | Successes (n) | Successes (%) | Difference | 90% CI Evaluation |
| Test | XXX | XXX | XX.X% | | |
| Reference | XXX | xxx | xx.x% | xx.x% | xx.x - xx.x |

#### **Superiority: modified Intent-to-Treat Population**

| | | Number of | Proportion of | |
|-----------|--------------|---------------|---------------|---------|
| Treatment | Number of | Treatment | Treatment | |
| Group | Subjects (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | xx.x% | |
| Test | XXX | XXX | xx.x% | x.xxxx |
| Reference | XXX | XXX | xx.x% | x.xxxx |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) exact test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)
Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)
Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

0453-01-01/

# T16.1.9.7.2 Summary of Supportive Analysis Results of Primary Efficacy Endpoint Proportion of Treatment Successes on the IGA (a score of 0 or 1 or 2) at the Week 12 Visit

| Equivalence: modified Intent-to-Treat Population | | | | | |
|---|---|---|---|---|---|
| | | | | Difference Between Treatments | |
| Treatment | Number of | Number of<br>Treatment | Proportion of<br>Treatment | | |
| Group | Subjects (N) | Successes (n) | Successes (%) | Difference | 90% CI Evaluation |
| Test | XXX | xxx | xx.x% | | |
| Reference | xxx | xxx | xx.x% | xx.x% | xx.x - xx.x |

#### **Superiority: Per-Protocol Population**

| | | Number of | <b>Proportion of</b> | |
|-----------|--------------|---------------|----------------------|---------|
| Treatment | Number of | Treatment | Treatment | |
| Group | Subjects (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | XX.X% | |
| Test | XXX | XXX | xx.x% | x.xxxx |
| Reference | XXX | XXX | xx.x% | X.XXXX |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) exact test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)
Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)
Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

0453-01-01/

# T16.1.9.8.1 Summary of Analysis Results of Secondary Efficacy Endpoint Proportion of Subjects with Disease Severity (a score of 0 or 1) on IGA at the Week 12 Visit

| <b>Equivalence: P</b> | Equivalence: Per-Protocol Population | | | | |
|---|---|---|---|---|---|
| | | | | Difference Between Treatments | |
| Treatment<br>Group | Number of<br>Subjects (N) | Number of<br>Treatment<br>Successes (n) | Proportion of Treatment Successes (%) | Difference | 90% CI Evaluation |
| Test | xxx | xxx | xx.x% | | |
| Reference | xxx | xxx | xx.x% | XX.X <sup>0</sup> / <sub>0</sub> | xx.x - xx.x |

#### **Superiority: modified Intent-to-Treat Population**

| | | Number of | <b>Proportion of</b> | |
|-----------|--------------|---------------|----------------------|---------|
| Treatment | Number of | Treatment | <b>Treatment</b> | |
| Group | Subjects (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | xx.x% | |
| Test | XXX | XXX | xx.x% | x.xxxx |
| Reference | XXX | XXX | xx.x% | x.xxxx |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) exact test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)
Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)
Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\\SAS\OU

\SAS\OUT

Created on: ddmmmyy hh:mm

0453-01-01/

# T16.1.9.8.2 Summary of Supportive Analysis Results of Secondary Efficacy Endpoint Proportion of Subjects with Disease Severity (a score of 0 or 1) on IGA at the Week 12 Visit

| Equivalence: modified Intent-to-Treat Population | | | | | |
|---|---|---|---|---|---|
| | | | | Difference Between Treatments | |
| | | Number of | <b>Proportion of</b> | | |
| Treatment | Number of | Treatment | Treatment | | |
| Group | Subjects (N) | Successes (n) | Successes (%) | Difference | 90% CI Evaluation |
| Test | xxx | xxx | xx.x% | | |
| Reference | xxx | xxx | xx.x% | xx.x% | xx.x - xx.x |

#### **Superiority: Per-Protocol Population**

| | | Number of | <b>Proportion of</b> | |
|-----------|--------------|---------------|----------------------|---------|
| Treatment | Number of | Treatment | Treatment | |
| Group | Subjects (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | xx.x% | |
| Test | XXX | XXX | xx.x% | x.xxxx |
| Reference | XXX | XXX | xx.x% | x.xxxx |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) exact test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

Protocol / 0453-01-01/

# T16.1.9.9.1 Summary of Analysis Results of Secondary Efficacy Endpoint Proportion of Subjects with Target Site Plaque Elevation, Scaling and Erythema Scores of Less Than or Equal to 1 on the PASI at the Week 12 Visit

| Equivalence: Per-Protocol Population | | | | | |
|---|---|---|---|---|---|
| | | | | Difference Between Treatments | |
| Treatment | Number of | Number of<br>Treatment | Proportion of<br>Treatment | | |
| Group | Subjects (N) | Successes (n) | Successes (%) | Difference | 90% CI Evaluation |
| Test | xxx | xxx | xx.x% | | |
| Reference | xxx | xxx | xx.x% | xx.x% | xx.x - xx.x |

# **Superiority: modified Intent-to-Treat Population**

| | | Number of | Proportion of | |
|-----------|--------------|---------------|---------------|---------|
| Treatment | Number of | Treatment | Treatment | |
| Group | Subjects (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | xx.x% | _ |
| Test | XXX | XXX | xx.x% | x.xxxx |
| Reference | XXX | XXX | xx.x% | X.XXXX |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) exact test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\\SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N



# T16.1.9.9.2 Summary of Supportive Analysis Results of Secondary Efficacy Endpoint Proportion of Subjects with Target Site Plaque Elevation, Scaling and Erythema Scores of Less Than or Equal to 1 on the PASI at the Week 12 Visit

| <b>Equivalence:</b> m | Equivalence: modified Intent-to-Treat Population | | | | |
|---|---|---|---|---|---|
| | | | | Difference Between Treatments | |
| Treatment | Number of | Number of<br>Treatment | Proportion of<br>Treatment | | |
| Group | Subjects (N) | Successes (n) | Successes (%) | Difference | 90% CI Evaluation |
| Test | xxx | xxx | xx.x% | | |
| Reference | xxx | xxx | xx.x% | xx.x% | xx.x - xx.x |

# **Superiority: Per-Protocol Population**

| | | Number of | <b>Proportion of</b> | |
|-----------|--------------|---------------|----------------------|---------|
| Treatment | Number of | Treatment | Treatment | |
| Group | Subjects (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | xx.x% | _ |
| Test | XXX | XXX | xx.x% | x.xxxx |
| Reference | XXX | XXX | xx.x% | X.XXXX |

The 90% confidence interval for the difference in proportions between test and reference was calculated using Yates' correction.

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) exact test, stratified by clinical site, at the 5% significance level using last observation carried forward (LOCF).

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\\SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

0453-01-01/

T16.1.9.10 Overall Summary of Adverse Events (Safety Population)

| Description | Test<br>N (%) | Reference<br>N (%) | Placebo<br>N (%) | Total<br>N (%) |
|---|---|---|---|---|
| Subjects Randomized | xxx | xxx | xxx | XXX |
| Subjects with at least one AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued study drug due to above AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AEs reported | XXX | XXX | XXX | xxx |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Suspected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Suspected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\

Created on: ddmmmyy hh:mm
## T16.1.9.11 Summary of Frequency of All Adverse Events by Body System (Safety Population)

| | Test (N = xxx) | | | Reference $(N = xxx)$ | | Placebo<br>(N = xxx) | | Fisher's |
|---|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Events | Subjects | Events | Subjects | Events | Subjects | P-value |
| Subject with at least one AE | Total | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | x.xxxx |
| Ear and labyrinth lisorders | Ear pain | XX | xx (xx.x%) | xx | xx (xx.x%) | XX | xx (xx.x%) | x.xxxx |
| | etc. | | | | | | | |

etc.

Comparison of treatment groups is with respect to the number of subjects with at least one occurrence of the AE.

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

T16.1.9.12 Summary of Frequency for AEs Occurring in at Least 5% of Subjects by Body System (Safety Population)

0453-01-01/ Protocol /

#### T16.1.9.13 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| | | | Test # Events (N=xx) | | | Reference # Events (N=xx) | | | Placebo<br># Events<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Total AEs | Total AEs | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Hypoacusis | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

etc.

N = Total number of events in each treatment group; Percentage is based on total number of events.

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\ \SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

T16.1.9.14 Summary of Frequency of All Adverse Events by Relationship (Safety Population)

| | | # I | Γest<br>Events<br>√=xx) | # F | erence<br>Events<br>V=xx) | # | Placebo<br>£ Events<br>(N=xx) |
|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Suspected | Not Suspected | Suspected | Not Suspected | Suspected | Not Suspected |
| Total AEs | Total AEs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Hypoacusis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | etc. | | | | | | |

etc.

N = Total number of events in each treatment group; Percentage is based on total number of events.

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

# T16.1.9.15 Summary of Frequency of Serious Adverse Events (Safety Population)

| | | Test | Reference | Placebo |
|---|---|---|---|---|
| Body System | MedDRA Term | # Events | # Events | # Events |
| Injury, poisoning and procedural complications | Alcohol poisoning | XX | XX | XX |

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

Protocol /

0453-01-01/

**T16.1.9.16 Summary of Application Site Reaction** (Safety Population)

| Signs and | | | Test | Reference | Placebo |
|---|---|---|---|---|---|
| Symptoms | Visit | Statistic | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ |
| Erythema | 1 | n | xxx | xxx | XXX |
| | | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | | Median | XX.X | XX.X | xx.x |
| | | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| | 2 | | | | |
| | 3 | | | | |
| | 4/ET | | | | |

Dryness

Burning/Stinging

Erosion

Edema

Pain

Itching

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

\SAS\OUT

Created on: ddmmmyy hh:mm

Protocol /

0453-01-01/

# T16.1.9.17 Summary of Frequency of Application Site Reaction (Safety Population)

| Signs and | | | Test | Reference | Placebo |
|-----------|-------|-----------|-------------|-------------|-------------|
| Symptoms | Visit | Statistic | (N = xxx) | (N = xxx) | (N = xxx) |
| Erythema | 1 | Absent | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Mild | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Moderate | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | | Severe | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |
| | 2 | | | | |
| | 3 | | | | |
| | 4/ET | | | | |

Dryness

Burning/Stinging

Erosion

Edema

Pain

Itching

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

\SAS\OUT

Created on: ddmmmyy hh:mm

## T16.1.9.18 Summary of Vital Signs (Safety Population)

| Vital Signs | Visit | Statistic | Test (N = xxx) | Reference $(N = xxx)$ | Placebo<br>(N = xxx) |
|---|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | 1 | n | XXX | XXX | XXX |
| | | $Mean \pm SD$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| | | Median | xxx.x | xxx.x | XXX.X |
| | | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| | 4/ET | | | | |

Diastolic Blood Pressure (mmHg)

Pulse Rate (beats/min)

Respiration Rate (breaths/min)

Temperature (F)

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\



Created on: ddmmmyy hh:mm

## L16.2.1 Listing of Discontinued Subjects

| Treatment | Subject | Discontinuation | |
|-----------|-----------|-------------------|------------|
| Group | Number | Reason | Population |
| Test | xx - xxxx | Withdrew Consent | Safety |
| | xx - xxxx | Lost to Follow-up | Safety |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

## L16.2.2 Listing of Protocol Deviations

| Treatment | Subject | | |
|-----------|-----------|-----------------------------------|------------|
| Group | Number | <b>Protocol Deviation Summary</b> | Population |
| Test | xx - xxxx | Outside Visit Window | Safety |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

## L16.2.3.1 Subjects Excluded from the Per-Protocol Population Data Set

| Treatment | Subject | Exclusion |
|-----------|-----------|-------------------------------------|
| Group | Number | Reason |
| Test | xx - xxxx | Subject did not meet IE criterion. |
| | xx - xxxx | Subject took prohibited medications |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

## L16.2.3.2 Subjects Excluded from the Modified Intent-to-Treat Data Set

| Treatment<br>Group | Subject<br>Number | Exclusion<br>Reason |
|---|---|---|
| Test | xx - xxxx | Subject did not have at least one post-randomization evaluation |
| | xx - xxxx | Subject did not have at least one post-randomization evaluation |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

## L16.2.4.1 Listing of Demographic Data

| Treatment | Subject | | | | | |
|---|---|---|---|---|---|---|
| Group | Number | Age | Sex | Ethnicity | Race | |
| Test | xx - xxxx | 30 | Female | Not Hispanic or Latino | Black or African American | , |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

#### L16.2.4.2 Listing of Medical History

| Treatment | Subject | | | | | |
|---|---|---|---|---|---|---|
| Group | Number | Category | Reported Term | <b>Onset Date</b> | <b>End Date</b> | Ongoing |
| Test | xx - xxxx | Gynecologic | Menopause | 2003 | 2003 | |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

0453-01-01/

## L16.2.4.3 Listing of Concomitant Medications

**Test: Tazarotene Cream 0.05%** 

| Subject | Medication/ | | | Start/End | | |
|---|---|---|---|---|---|---|
| Number | Therapy Name | Dosage | Frequency | Route | Date | Indication |
| xx - xxxx | LISINOPRIL | 20 MG | QD | PO | yyyy-mm-dd/ | HYPERTENSION |

Note to programmer: table will continue for reference and placebo group

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

\SAS\OUT

Created on: ddmmmyy hh:mm

## L16.2.5.1 Listing of Visit Date Information

| Treatment | Subject | Inform Consent | | | | Visit 4 or |
|---|---|---|---|---|---|---|
| Group | Number | Date | Visit 1 | Visit 2 | Visit 3 | <b>Early Termination</b> |
| Test | xx - xxxx | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd |

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT Created on: ddmmmyy hh:mm

Protocol /

0453-01-01/

## L16.2.5.2 Listing of Drug Administration

| Treatment | Subject | Date of | Date of | Total Doses | Dosing |
|---|---|---|---|---|---|
| Group | Number | First Dose | Last Dose | Applied | Compliance (%) |
| Test | xx - xxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX.X |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

\SAS\OUT

Created on: ddmmmyy hh:mm

#### L16.2.6.1 Listing of Investigator Global Assessment (IGA)

| Treatment<br>Group | Subject<br>Number | Visit 1 | Visit 2 | Visit 3 | Visit 4 or<br>Early Termination | Treatment<br>Success* | Treatment Success** |
|---|---|---|---|---|---|---|---|
| Test | xx - xxxx | 4 | 4 | 3 | 0 | Yes | Yes |
| | xx - xxxx | 4 | 4 | 3 | 2 | Yes | No |
| | xx - xxxx | 4 | 4 | 3 | 3 | No | No |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial \SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

<sup>\*</sup>Treatment Success: defined as none, minimal or mild disease, a score of 0, 1 or 2 within the treatment area on the IGA at the Week 12 visit (Day  $85 \pm 4$  days, End of Study).

<sup>\*\*</sup>Treatment Success: defined as subjects with disease severity at the Week 12 visit (Day 85 ± 4 days, End of Study) consistent with none or minimal, a score of 0 or 1, within the treatment area on the IGA

Protocol /

0453-01-01/

L16.2.6.2 Listing of Psoriasis Area Severity Index (PASI) at the Target Lesion Site

| Treatment<br>Group | Subject<br>Number | Visit | Scaling | Erythema | Plaque<br>Elevation | PASI<br>Score | Clinical<br>Success |
|---|---|---|---|---|---|---|---|
| Test | xx - xxxx | 1 | 2 | 3 | 1 | 6 | |
| | | 2 | 2 | 3 | 1 | 6 | |
| | | 3 | 1 | 2 | 1 | 4 | |
| | | 4/ET | 1 | 1 | 0 | 2 | Yes |
| | xx - xxxx | 1 | 2 | 3 | 1 | 6 | |
| | | 2 | 2 | 3 | 1 | 6 | |
| | | 3 | 1 | 2 | 1 | 4 | |
| | | 4/ET | 1 | 2 | 0 | 3 | No |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

## L16.2.6.3 Listing of Dermatological Examination

| | | | | | Location | Target Lesion _ | | % BSA A | ffected | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject<br>Number | Height (cm) | Weight<br>(kg) | BSA<br>(m^^2) | of the<br>Target Lesion | Area | V1 | V2 | V3 | V4/ET |
| Test | xx - xxxx | XXX | xxx.x | XXX.X | Head front | XXX.X | xxx.x | xxx.x | xxx.x | XXX.X |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

## L16.2.7.1 Listing of Adverse Events by Treatment Group

**Test: Tazarotene Cream 0.05%** 

| Subject | Body System/ | | TX Start /End | | Relationship<br>to Investigational | | Action Taken with<br>Investigational<br>Drug / | |
|---|---|---|---|---|---|---|---|---|
| Number | AE Term | Area | Date | Severity | Drug | Outcome | Other Action Taken | SAE? |
| XX - XXXX | Nervous system disorders/ headache/<br>Headache | No | yyyy-mm-dd /<br>yyyy-mm-dd | Mild | Not Suspected | Recovered | Drug withdrawn/ None | No |

Note to programmer: table will continue for reference and placebo group

Path: L:\Studies\_Sas\_Codes\Clinical Trial\\SAS\OUT Created on: ddmmmyy hh:mm Page 1 of N

## L16.2.7.2 Listing of Application Site Reactions

| | | | | Burning | | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Visit | Erythema | Dryness | /Stinging | Erosion | Edema | Pain | Itching |
| Test | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |
| | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |
| | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |
| | 4/ET | 0 | 0 | 0 | 1 | 0 | 0 | 2 |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)

Reference: TAZORAC (tazarotene) Cream, 0.05% (Allergan, Inc.)

Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\



Created on: ddmmmyy hh:mm

## L16.2.8.1 Listing of Pregnancy Test Results

| Treatment | Subject | | | | Visit 4 or |
|---|---|---|---|---|---|
| Group | Number | Visit 1 | Visit 2 | Visit 3 | <b>Early Termination</b> |
| Test | xx - xxxx | Negative | Negative | Negative | Negative |

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.)
Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.)
Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies\_Sas\_Codes\Clinical Trial\

\SAS\OUT

Created on: ddmmmyy hh:mm

#### L16.2.8.2 Listing of Vital Signs

| Treatment<br>Group | Subject<br>Number | Visit | Systolic BP (mmHg) | Diastolic BP<br>(mmHg) | Pulse Rate<br>(beats/min ) | Respiration Rate (breaths/min) | Temperature<br>(F) |
|---|---|---|---|---|---|---|---|
| Test | xx - xxxx | 1 | 120 | 70 | 84 | 18 | 98.6 |
| | | 4/ET | 140 | 80 | 74 | 18 | 97 |

xx - xxxx

Reference

Placebo

Test: Tazarotene Cream 0.05% (Fougera Pharmaceuticals Inc.) Reference: TAZORAC® (tazarotene) Cream, 0.05% (Allergan, Inc.) Placebo: Placebo (vehicle) Cream (Fougera Pharmaceuticals Inc.)

Path: L:\Studies Sas Codes\Clinical Trial\\SAS\OUT

Created on: ddmmmyy hh:mm

#### STATISTICAL ANALYSIS PLAN

**Tazarotene Cream 0.05%** 

Protocol /

0453-01-01/

## APPENDIX A: Investigator's Global Assessment of Disease Severity

| Score | Grade | Definition |
|---|---|---|
| 0 | None | No plaque elevation above normal skin level; may have residual non-<br>erythematous discoloration; no psoriatic scale; no erythema |
| 1 | Minimal | Essentially flat with possible trace elevation; faint erythema; no psoriatic scale |
| 2 | Mild | Slight but definite elevation of plaque above normal skin level; may have up to moderate erythema (red coloration); fine scales with some lesions partially covered |
| 3 | Moderate | Moderate elevation with rounded or sloped edges to plaque; moderate erythema (red coloration); somewhat coarse scales with most lesions partially covered |
| 4 | Severe | Marked elevation with hard, sharp edges to plaque; severe erythema (very red coloration); coarse, thick scales with virtually all lesions covered and a rough surface |
| 5 | Very<br>Severe | Very marked elevation with very hard, sharp edges to plaque; very severe erythema (extreme red coloration); very coarse, thick scales with all lesions covered and a very rough surface |

To be eligible for participation in the study a subject must have a Baseline IGA score of 3, 4 or 5.

A subject shall be considered a "treatment success" if he/she has an IGA score of 0, 1 or 2 within the treatment area at the Week 12 visit.

#### STATISTICAL ANALYSIS PLAN

**Tazarotene Cream 0.05%** 

Protocol /

0453-01-01/

## APPENDIX B: Psoriasis Area Severity Index at the Target Lesion Site

| Score | Grade | Erythema | Scaling | Plaque Elevation |
|---|---|---|---|---|
| 0 | Clear | No evidence of | No evidence of | No evidence of plaques |
| | | erythema | scaling | above normal skin level |
| 1 | Almost | Pink discoloration, | Occasional fine | Slight, just discernible |
| | Clear | minimal erythema | scales hardly | elevation above normal |
| | | | noticeable | skin level |
| 2 | Mild | Light red coloration | Slight but definite | Discernible elevation |
| | | | roughness, fine scale | above normal skin level |
| | | | present, no cracking | upon examination, but |
| | | | | not pronounced |
| 3 | Moderate | Moderate redness, | Moderate roughness, | Definite plaque |
| | | but not dark | somewhat coarse | formation with |
| | | | scaling | rounded/sloped edges to |
| | | | | plaque |
| 4 | Severe | Dark red coloration | Marked roughness, | Marked elevation with |
| | | | coarse/thick scaling, | hard, distinct edges to |
| | | | cracking may be | plaque |
| | | | evident | |
| 5 | Very | Very dark red | Very thick scales | Very marked elevation, |
| | Severe | coloration with | covering extensive | very hard and sharp |
| | | induration present | area, severe | edges to plaque |
| | | | cracking/fissures may | |
| | | | be evident | |

To be eligible for participation in the study a subject must have a minimum plaque elevation of at least moderate severity (score  $\geq 3$ ) at the target lesion site. The most severe lesion at Baseline should be identified as the target lesion.

#### STATISTICAL ANALYSIS PLAN

#### **Tazarotene Cream 0.05%**

Protocol /

0453-01-01/

## **APPENDIX C: Application Site Reactions**

The following application site reactions will be evaluated at each visit based on the scale provided below:

#### Signs and Symptoms:

Erythema

Dryness

Burning/Stinging

**Erosion** 

Edema

Pain

Itching

## **Grading Scale:**

| Severity | <u>Grade</u> |
|----------|--------------------------------|
| Absent | 0 |
| Mild | 1 (slight, barely perceptible) |
| Moderate | 2 (distinct presence) |
| Severe | 3 (marked, intense) |